CLINICAL TRIAL: NCT00888914
Title: A Phase 2, Double-Blind, Randomized, Parallel-Group, Controlled, Dose-Ranging, Multi-Center Study to Evaluate the Safety and Efficacy of RT001, a Botulinum Toxin Type A Topical Gel, to Treat Moderate to Severe Lateral Canthal Lines in Adults.
Brief Title: Safety and Efficacy Study of RT001 to Treat Moderate to Severe Lateral Canthal Lines
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RT001-CL006LCL
Record Dates: First submitted 2009-04-24; First posted 2009-04-28 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-10

CONDITIONS: Lateral Canthal Lines; Crow's Feet; Facial Wrinkles
Keywords: Lateral Canthal Lines; Crow's Feet; Facial Wrinkles
MeSH Terms: interventions — RT001

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Dose A (Active Comparator): RT001 Dose A; Active Comparator
  Interventions: Drug: RT001
- Dose B (Active Comparator): RT001 Dose B; Active Comparator
  Interventions: Drug: RT001
- Dose C (Active Comparator): RT001 Dose C; Active Comparator
  Interventions: Drug: RT001
- Dose D (Active Comparator): RT001 Dose D; Active Comparator
  Interventions: Drug: RT001
- Dose E (Placebo Comparator): RT001 Dose E; Vehicle Comparator
  Interventions: Other: Vehicle Comparator

INTERVENTIONS:
Drug: RT001 — RT001
  Arms: Dose B
Drug: RT001 — RT001
  Arms: Dose A
Drug: RT001 — RT001
  Arms: Dose C
Drug: RT001 — RT001
  Arms: Dose D
Other: Vehicle Comparator — Vehicle Comparator
  Arms: Dose E

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of RT001 to treat moderate to severe lateral canthal lines in adults.

DETAILED DESCRIPTION:
This multi-center study evaluates the safety and efficacy of four different doses of RT001 compared to vehicle applied as a single, bilateral topical application in at least 60 subjects with moderate to severe lateral canthal lines. Subjects will be randomized to one of the five treatment groups in a 1:1:1:1:1 ratio. Follow-up visits are scheduled through 28 days post-treatment. The safety and efficacy of Cohort 1 (through the Day 14 visit) will be assessed prior to the decision to enroll subjects into Cohort 2 if additional doses or treatment regimens need to be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Female or male; 30 to 55 years of age
* Bilateral lateral canthal lines rated as moderate or advanced
* Willing to refrain from receiving facial fillers, laser treatments, use of any product that affects remodeling or a product that may cause an active dermal response in the treatment area beginning at Screening through End of Study
* Women of childbearing potential must be practicing and willing to continue to use an effective method of birth control during the course of the study

Exclusion Criteria:

* Muscle weakness or paralysis in the area receiving study treatment
* Active skin disease or irritation at the treatment areas
* Undergone any procedures that may affect the lateral canthal region during the past 12 months prior to Screening
* Previous treatment with botulinum toxin (any serotype) in the head or neck area within 9 months prior to Baseline (Day 0)
* Use of a topical steroid on either of the treatment areas or use of medications that suppress the immune system 30 days prior to Screening and continuing through End of Study (Day 28)
* Any abnormality on the electrocardiogram (ECG) at Screening or any history of clinically significant arrhythmia, unstable angina, myocardial infarction or congestive heart failure

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2008-11; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The number of subjects classified as exhibiting improvement via the Investigator Global Assessment at Smile from Baseline (Day 0) to End of Study (Day 28) | Day 28

SECONDARY OUTCOMES:
The number of subjects classified as exhibiting improvement via the Investigator Global Assessment at Rest from Baseline (Day 0) to End of Study (Day 28) | Day 28
Incidence of treatment-emergent AEs | Day 28

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Richard G. Glogau, MD, San Francisco, California
  - Head and Neck Surgical Group, New York, New York
  - Aesthetic Plastic Surgery, New York, New York
  - Dermatology Surgery and Laser Center, White Plains, New York